CLINICAL TRIAL: NCT07175467
Title: Development and Implementation of a Multi-Skill, Haptic-Supported Virtual Reality Simulation for Nursing Students
Brief Title: Development and Implementation Haptic VR Simulation
Acronym: VR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, özlem doğu, Project Manager, Sakarya University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: E-61923333-050.99-285112
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Nursing; Skill Performance; Virtual Reality; Simulation-based Training
Keywords: nursing; virtual reality; skills training; clinical decision making; haptic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haptic-assisted virtual reality (Experimental): The haptic-assisted virtual reality simulation developed for the intervention group will enable them to practice nursing skills.
  Interventions: Other: Haptic-asissted virtual simulation
- Control (No Intervention): Classic nursing skills education with task trainer in the nursing skills laboratory.

INTERVENTIONS:
Other: Haptic-asissted virtual simulation — The virtual reality application will be developed using the Unity game engine. The VR simulation environment, which will progress through scenarios, will include taking vital signs, performing aspiration, performing a nasogastric catheterization, oxygen therapy, performing physical examinations, and performing subcutaneous injections.
  Arms: Haptic-assisted virtual reality

SUMMARY:
The goal of this experimental study is to increase objectivity in clinical decision-making and skill assessment of nursing students by using haptic-assisted virtual reality simulation, unlike imported products used in nursing education.

Hypotheses:

H1: There is a difference between the total psychomotor skill levels of the intervention and control group students in all relevant skill applications.

H2: There is a difference between the clinical decision-making score averages of the intervention and control group students.

Researchers will compare the effects of haptic-assisted virtual simulation training on psychomotor skill levels and clinical decision-making scores in the intervention and control groups.

Participants will:

* Students who have agreed to participate in the study,
* Students taking the Fundamentals of Nursing course for the first time,
* Students with no prior simulation experience

ELIGIBILITY:
Inclusion Criteria:

* Students who have agreed to participate in the study,
* Students taking the Fundamentals of Nursing course for the first time,
* Students with no prior simulation experience

Exclusion Criteria:

* Students who do not meet the inclusion criteria,
* Students who do not complete the data collection forms in full,
* Students who are retaking the Fundamentals of Nursing course will be excluded from the study.
* Students who do not participate in the virtual reality application or laboratory application to be implemented during the study period, who are absent, or who wish to withdraw from the study will be excluded from the study during the follow-up period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Decision Making, Self-Confidence, and Anxiety Assessment in Nursing | 1 month
  This scale assesses nursing students' anxiety and self-confidence levels in clinical decision-making. Separate scores are obtained for self-confidence and anxiety from the scale, which consists of a total of 27 questions. Both the self-confidence and anxiety sections of the scale have three subscales: "Using resources to obtain information and listening carefully (13 questions)", "Using available information to identify the problem (7 questions)", and "Knowing and taking action (7 questions)". Higher scores on self-confidence and its subdimensions indicate increased levels of self-confidence in clinical decision-making among students. Low scores on the anxiety section and its subdimensions indicate low levels of anxiety in clinical decision-making. It is a six-point Likert-type scale. The lowest possible score on the self-confidence and anxiety sections is 27, and the highest possible score is 162.
Knowledge Test | 1 month
  The Knowledge Test, prepared in line with the literature, consists of 20 questions. Each question will be scored with "1" point for a correct answer and "0" points for an incorrect answer. Questions covering all skill applications will be scored out of 100, with the total number of correct answers completing the score. The form was evaluated by ten experts in the field of Nursing Fundamentals outside of the study and finalized. The purpose of the expert opinion is to examine the items according to criteria such as whether the test measures behavior according to its structure, its comprehensibility in terms of language, whether there are scientific errors, grammatical errors, and the suitability of the items for the group to be applied to, and to make the necessary corrections.
Performance evaluation | 1 month
  The performance report, which awards points out of 100, will include scoring for nursing interventions. Performance report scores range from 0 to 100; minimum score "0", maximum score "100". The performance report applied with the task trainer has been created to be identical to the virtual patient simulation performance report, and OSCE steps have been defined. The performance forms created will be evaluated by the researcher during the student's application. All students (intervention and control groups) will use the application at least once within the scope of the study. For the success assessment in the applications, the cutoff score is considered as follows: 50.00-59.99 is passing, 60.00-69.99 is average, 70.00-84.99 is good, and 85.00-100 is excellent. A higher score indicates higher performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Faculty of Health Sciences, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
There are plans to make the IPD and related data dictionaries available for use. Researchers may share the data upon request after the study is published.
Supporting Information: SAP
Time Frame: After the study is published, researchers may share the data for a period of three years upon request.
Access Criteria: Researchers in the field of nursing may contact the researchers of this study to request the data.

REFERENCES:
- [Background] White KA. Development and validation of a tool to measure self-confidence and anxiety in nursing students during clinical decision making. J Nurs Educ. 2014 Jan 1;53(1):14-22. doi: 10.3928/01484834-20131118-05. Epub 2013 Nov 18. PMID 24256004
- [Background] Park S, Hur HK, Chung C. Learning effects of virtual versus high-fidelity simulations in nursing students: a crossover comparison. BMC Nurs. 2022 Apr 27;21(1):100. doi: 10.1186/s12912-022-00878-2. PMID 35473614
- [Background] Butt, A. L., Kardong-Edgren, S., & Ellertson, A. (2018). Using game-based virtual reality with haptics for skill acquisition. Clinical Simulation in Nursing, 16, 25-32.
- [Background] Sundler AJ, Pettersson A, Berglund M. Undergraduate nursing students' experiences when examining nursing skills in clinical simulation laboratories with high-fidelity patient simulators: A phenomenological research study. Nurse Educ Today. 2015 Dec;35(12):1257-61. doi: 10.1016/j.nedt.2015.04.008. Epub 2015 Apr 25. PMID 25943280
- [Background] Sanders, D. (2010). Comparing ability to complete simple tele-operated rescue or maintenance mobile-robot tasks with and without a sensor system. Sensor Review, 30(1), 40-50.
- [Background] Kim, S. Y., Han, H. G., Kim, J. W., Lee, S., & Kim, T. W. (2017). A hand gesture recognition sensor using reflected impulses. IEEE Sensors Journal, 17(10), 2975-2976.